CLINICAL TRIAL: NCT02886819
Title: Whole-body Vibration Induces a Short or Long Latency Muscular Reflex Depending on Vibration Intensity
Brief Title: Whole-body Vibration Induces a Short or Long Latency Muscular Reflex
Acronym: WBV-IMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BEAH FTR-11
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Effects of Vibration
Keywords: Whole body vibration; Tonic vibration reflex; Bone myoregulation reflex
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WBV group (Experimental): whole-body vibration (WBV) group
  Interventions: Other: vibration

INTERVENTIONS:
Other: vibration — Whole body vibration
  Other Names: Whole body vibration

SUMMARY:
Aim: Hypothesis of this study was that WBV activates different receptors or reflex pathways depend on vibration intensity. Aim of this study was to test this hypothesis.

Methods: This study was conducted on 11 healthy adults. WBV was applied at various frequencies and amplitudes. The right soleus T-reflex latency was determined before and during WBV. WBV-IMR latency of the right soleus was determined using two different vibration intensity: weak vibration and powerful vibration. T-reflex latency and WBV-IMR latency were determined by using cumulated average method.

DETAILED DESCRIPTION:
Aim: Whole-body vibration (WBV) induces a reflex response in muscles. The physiological mechanisms underlying this reflex have been explained by activating muscle spindles (stretch-induced reflex) or osteocytes (bone myoregulation reflex). WBV-induced muscular reflex (WBV-IMR) latency was reported to be significantly longer than latency of T-reflex as a stretch-induced reflex or nearly equal to T-reflex latency in the literatures. Hypothesis of this study was that WBV activates different receptors or reflex pathways depend on vibration intensity. Aim of this study was to test this hypothesis.

Methods: 2.1. Participants

Eleven young, healthy and right hand dominant male adult volunteers were included in this study. The mean age of the participants was 25.4 ± 4.7 years, mean body height was 176.5 ± 6.7 cm and mean body weight was 77.8 ± 13.8 kg. All volunteers gave written informed consent to the experimental procedures, which were in accordance with the Declaration of Helsinki and were approved by the local ethics committee (Yeditepe University Medical Faculty Clinical Research Evaluation Committee, Istanbul; 2016/564 ).

2.2. Procedure Prior to the induction of WBV, control T-reflex recordings were elicited and then the participants completed a 15-s trial WBV protocol to familiarize themselves with the procedure. Following the control T-reflex recordings, the trial protocol and a 15-s rest, the participants received three set of WBV and T-reflex stimuli during WBV. A weak vibration was applied in the first set. In next sets, a moderate and strong vibration were applied, respectively. Vibration characteristics of three sets was given in Table 1. A WBV set consisted of four vibration periods, each lasting for 60 s, with 5-s rest intervals between periods. Within each set, WBV frequencies of 25, 29, 33, and 37 Hz were delivered The surface electromyography (SEMG) and accelerometer data were obtained while the participants stood upright on the vibration platform with the knees in extension. The participants were barefooted and stood directly on the vibration platform. The whole plate oscillated with a linear movement upward and downward. Two WBV devices (Power-Plate®Pro5, PowerPlate® International, Ltd. London, UK) were used in the present study. One of them was used for applying the moderate and strong vibration. The other WBV device was modified to attenuate vibration intensity and used for applying the weak vibration.

2.3. Data Recordings The recordings of both T-reflex and WBV-IMR were acquired using SEMG. The Ag/AgCl electrodes (KENDALL®Covidien) with a disc radius of 10 mm were placed 20 mm apart on the right soleus muscle belly on shaved skin that had been cleaned with alcohol in accordance with the recommendations of the Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) project (Hermens et al., 2000). The ground electrode was placed on the lateral malleolus. The sampling frequency was selected as 10 kHz.

A very light (2.9 g) triaxial MEMS piezoaccelerometer (LIS344ALH, full-scale of ± 6 g, linear accelerometer, ECOPACK®) was taped to the participant's right Achilles tendon to determine the timing of the onset of the mechanical stimulus for the T-reflex and to measure stroke intensity of reflex hammer to Achilles tendon (Achilles accelerometer). Similar accelerometers fixed to the WBV platforms to determine the timing of the onset of the mechanical stimulus for the WBV-IMR (platform accelerometers). Acceleration unit used in this study was m/s2.

A custom-made reflex hammer tapped the right Achilles tendon just caudal to the accelerometer with a force of about 19.6 N. Before vibration and in each vibration session, the Achilles tendon was tapped ten times with approximately 3-s intervals between taps.

2.4.Data processing SEMG and accelerometer data were recorded using a PowerLAB® data acquisition system (ADInstruments, Oxford, United Kingdom) and the data were analyzed offline using the LabChart7® (ver 7.3.7, ADInstruments, Oxford, United Kingdom) software. A sampling frequency of 10 kHz was used. All accelerometer recordings were filtered with high-pass filter set at 5 Hz. All EMG recordings were filtered using a band pass filter from 60 to 500 Hz.

The maximum peak-to-peak (PPmax) amplitudes of T-reflex were determined for each vibration session. The amplitude of WBV-IMR was expressed as the Root Mean Square (RMS). The PPmax amplitude of T-reflex and RMS amplitude of WBV-IMR recorded during the strong WBV were used to normalize of the PPmax amplitude of T-reflex and RMS amplitude of WBV-IMR recorded before WBV or during weak and moderate WBV.

In the present study, reflex latency was defined as the time between the onset of the mechanical stimulus and the onset of the EMG spike on the cumulated average trace, both of which were determined using the cumulative average method, as previously described (Karacan et al). The positive peaks of the rectified EMG data were used as a trigger to average the accelerometer data and the rectified EMG data. The point on the cumulative average trace of the platform accelerometer data where the standard error (SE) was the lowest was considered the stimulus onset point. The point on the cumulative average trace of the rectified EMG data where the SE was lowest was considered the point of onset for the EMG spike. The mean height of young adult males in country (175 cm) was used to normalize of the T-reflex and WBV-IMR latencies (Cidem et al).

2.5. Precautions for voluntary muscle contractions and motion artifacts Five measures were taken: 1) the participants were asked to use the handles of the WBV device to secure their balance. The sense of balance may impair during WBV. Therefore muscles may be activated to restore balance during WBV, 2) Before WBV trials, participants were asked to relax and not to make voluntary contractions in their lower extremity muscles. This instruction was provided with verbal feedback given by the researcher who monitored the SEMG recordings from the screen. If the RMS amplitude of EMG was lower than five microvolts during this intruction, it was accepted that muscle relaxation was accomplished by participant, 3) a trial protocol was applied to familiarize vibration, 4) all cables were carefully taped to the skin to minimize motion artifacts, 5) all EMG recordings were filtered to avoid WBV induced movement artifacts (Sebik et al., 2013).

2.6. Statistical analysis The normal distribution of the data was confirmed using the Kolmogorov-Smirnov test. Continuous variables were summarized as arithmetic mean and standard deviation (SD).

The paired sample t-test was used to analyze the statistical difference in the amplitude of WBV-IMR between weak and moderate WBV. General linear model repeated measures test was used to compare in the T-reflex latencies, WBV-IMR latencies or PPmax amplitude of T-reflex among the sessions. The alpha (α) threshold was chosen as 0.05. The Bonferroni test was applied for pair-wise comparisons (PostHoc analyses). Using a Bonferroni (a significance level for each pair-wise comparisons is α/m, m is the number of pair-wise comparisons), results with a p value ≤ 0.017 were considered significant. Confidence interval (CI), mean, and standard error (SE) were calculated for all data. When comparing means of two data sets, if ±95% CI of one data set included the mean of another data set, it was established that there is no statistical difference between the means of two data sets. The data management software package used was PASW statistics (formerly SPSS Statistics) for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Right-handed men

Exclusion Criteria:

* Bone, muscle/tendon, joint, vascular, dermatologic diseases in lower extremities and spine
* Medication that could affect the musculoskeletal system
* Postural abnormalities (scoliosis, kyphosis, etc)
* Systemic diseases

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
latency of reflex muscle activity | 1 month

IPD SHARING:
Plan to Share IPD: No